CLINICAL TRIAL: NCT06479135
Title: A Phase 3, Randomized, Double-blind, Add-on Study Evaluating the Safety and Efficacy of Navtemadlin Plus Ruxolitinib vs Placebo Plus Ruxolitinib in JAK Inhibitor-Naïve Patients With Myelofibrosis Who Have a Suboptimal Response to Ruxolitinib
Brief Title: Study of Navtemadlin add-on to Ruxolitinib in JAK Inhibitor-Naïve Patients With Myelofibrosis Who Have a Suboptimal Response to Ruxolitinib
Acronym: POIESIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRT-232-115
Record Dates: First submitted 2024-06-21; First posted 2024-06-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-10

CONDITIONS: Myelofibrosis; Post-PV MF; Post-ET Myelofibrosis; Primary Myelofibrosis; MF
Keywords: Navtemadlin; KRT-232; Ruxolitinib; POIESIS; TP53; Suboptimal response; Sub-optimal response
MeSH Terms: conditions — Primary Myelofibrosis | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Navtemadlin administered orally once daily on Days 1-7, off treatment on Days 8-28, in 28-day treatment cycles. Ruxolitinib administered orally twice a day.
  Interventions: Drug: Navtemadlin; Drug: Ruxolitinib
- Arm 2 (Active Comparator): Navtemadlin placebo administered orally once daily on Days 1-7, off treatment on Days 8-28, in 28-day treatment cycles. Ruxolitinib administered orally twice a day.
  Interventions: Drug: Navtemadlin placebo; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Navtemadlin — Navtemadlin is an investigational MDM2 inhibitor
  Other Names: KRT-232
  Arms: Arm 1
Drug: Navtemadlin placebo — Navtemadlin placebo
  Other Names: KRT-232
  Arms: Arm 2
Drug: Ruxolitinib — Ruxolitinib is a janus kinase 1/2 inhibitor
  Other Names: Jakafi; Jakavi

SUMMARY:
This clinical trial is evaluating whether addition of navtemadlin to ruxolitinib treatment will provide more clinical benefit than ruxolitinib alone for patients with Myelofibrosis who have a suboptimal response to ruxolitinib treatment alone.

Subjects will start by receiving ruxolitinib alone in the run-in period. Those who demostrate a suboptimal response from ruxolitinib alone will then be randomized 2:1 to receive navtemadlin or navtemadlin placebo as add-on treatment to their ongoing ruxolitinib. Randomized means that subjects will be assigned to a group by chance, like a flip of a coin. The study is blinded, meaning the subjects, doctors, central endpoint assessors and sponsor will not know which add on treatment (navtemadlin or navtemadlin placebo) the subject is receiving.

ELIGIBILITY:
Inclusion Criteria for Ruxolitinib Alone Period:

* Confirmed diagnosis of PMF, post-PV MF, or post-ET MF, as assessed by the treating physician according to the World Health Organization (WHO) criteria
* High, Intermediate-1, Intermediate-2 risk category International Prognosis System Score (IPSS)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* JAK-inhibitor treatment naive

Exclusion Criteria for Ruxolitinib Alone Period:

* Prior Splenectomy
* Splenic irradiation within 3 months prior to the first dose
* Prior BCL-XL, BET, MDM2, PI3K, PIM, or XPO1 inhibitors therapy or p53-directed therapy
* Eligible for Bone Marrow Transplant
* Peripheral blood or bone marrow blast count ≥ 10 percent

Inclusion Criteria for Randomized Period:

* PMF, post-PV MF, or post-ET MF that is TP53WT as assessed by central testing
* ECOG performance status of 0 to 2
* Treatment with a stable dose of ruxolitinib
* Suboptimal response to run-in ruxolitinib treatment

Exclusion Criteria for Randomized Period:

* Elevated white blood cell count that doubles (or more) during ruxolitinib treatment and exceeds 50 × 10^9/L
* Peripheral blood or bone marrow blast count ≥ 10 percent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare spleen volume reduction (SVR35) between Arm 1 and Arm 2 | 24 weeks
  The proportion of subjects in each arm with SVR35 by MRI/CT scan (central review) 24 weeks after start of the randomized period
To compare total symptom score reduction (TSS50) between Arm 1 and Arm 2 | 24 weeks
  The proportion of subjects in each arm with a TSS50 by the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 24 weeks after start of the randomized period

SECONDARY OUTCOMES:
To compare time to progression between Arm 1 and Arm 2 | Up to 8 years
  Time to progression or death from any cause in subjects randomized to each arm
To compare overall survival (OS) between Arm 1 and Arm 2 | Up to 8 years
  Time to death from any cause in subjects randomized to each arm

CONTACTS AND LOCATIONS:
Locations (215):
- United States (58):
  - UAB Hospital, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology Clinic - Los Angeles, Los Angeles, California
  - Scripps Health, Prebys Cancer Center, San Diego, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - MedStar Georgetown University Hospital, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mission Cancer + Blood, Des Moines, Iowa
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Cancer Institute - Brigitte Harris Cancer Pavilion, Detroit, Michigan
  - Nebraska Hematology - Oncology, P.C., Lincoln, Nebraska
  - Mohtaseb Cancer Center and Blood Disorders, Henderson, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Cayuga Cancer Center, Ithaca, New York
  - Northwell Health, R.J. Zuckerberg Cancer Center, Lake Success, New York
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - Medical University of South Carolina (MUSC), Charleston, North Carolina
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Independence Family Health Center - Cleveland Clinic, Independence, Ohio
  - Hillcrest Hospital - Cleveland Clinic, Mayfield Heights, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT - SouthWestern, Dallas, Texas
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Virginia Oncology Associates - Virginia Beach, Virginia Beach, Virginia
  - Fred Hutchinson Cancer Centre, Seattle, Washington
  - Northwest Medical Specialties, PLLC - Tacoma, Tacoma, Washington
  - Sheboygan Cancer & Blood Specialists, Sheboygan, Wisconsin
- Australia (11):
  - Royal Hobart Hospital (RHH), Hobart, Tasmania
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Monash Medical Center Clayton, Clayton
  - Townsville University Hospital, Douglas
  - Gosford Hospital, Gosford
  - St George Hospital, Kogarah
  - The Royal Melbourne Hospital - Peter MacCallum Cancer Center, Melbourne
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
  - Calvary Mater Newcastle Hospital, Waratah
- Austria (7):
  - University Hospital Graz, Department of Internal Medicine, Graz
  - Medical University Innsbruck, Department of Internal Medicine V (Hematology and Oncology), Innsbruck
  - Regional Hospital Hochsteiermark - Leoben, Department of Internal Medicine, Department of Hematology and Oncology, Leoben
  - Ordensklinikum Linz GmbH Elisabethinen Hospital, Department of Internal Medicine I - Hemato-Oncology, Linz
  - Kepler University Hospital GmbH, Med Campus 3, University Clinic for Hematology and Internal Oncology, Linz
  - Medical University Vienna, Vienna
  - Hospital Ottakring, Department of Internal Medicine I, Vienna
- Belgium (5):
  - Antwerp Hospital Network (ZNA) Cadix, Antwerp
  - University Hospitals Leuven, Campus Gasthuisberg, Leuven
  - University Hospital Center Sart-Tilman, Liège
  - General Hospital Delta, Roeselare
  - UCL Mont-Godinne University Hospitals, Yvoir
- Croatia (7):
  - Clinical Hospital Centre Rijeka, Rijeka
  - University Hospital of Split, Split
  - General Hospital of Sibenik-Knin County, Šibenik
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Merkur, Zagreb
  - Solmed Clinic, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (5):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Ostrava, Ostrava
  - University Hospital Kralovske Vinohrady, Prague
  - Institute of Hematology and Blood Transfusion, Prague
- France (14):
  - Saint-Louis Hospital, Department of Adult Hematology, Paris, Paris
  - Amiens Picardie University Hospital - South, Amiens
  - Angers University Hospital Center, Angers
  - Lille Regional University Hospital Center, Lille
  - South Lyon Hospital Center, Lyon
  - Leon Berard Center, Lyon
  - Nantes University Hospital Center - Hotel Dieu Hospital, Nantes
  - Archet 1 and 2 hospital, Nice
  - Nimes University Hospital Center, Department of Clinical Hematology and Medical Oncology, Nîmes
  - Bordeaux University Hospital, Pessac
  - University Hospital Center of Poitiers, Poitiers
  - Strasbourg Europe Institut of Cancerology, Strasbourg
  - University Hospital of Toulouse, IUCT-Oncopole, Toulouse
  - Tours Regional University Hospital Center, Tours
- Georgia (6):
  - JSC Vian, Kutaisi
  - JSC German Hospital, Tbilisi
  - LEPL The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Caucasus Medical Centre LLC, Tbilisi
- Germany (14):
  - Marien Hospital Duesseldorf GmbH, Düsseldorf
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Halle (Saale), Halle
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Jena, Jena
  - University Hospital Schleswig-Holstein, Kiel
  - MVZ Mitte Am Johannisplatz, Leipzig
  - Hospital Rechts der Isar, Munich
  - Staufer Schwaebisch Gmuend Hospital, Mutlangen
  - Hospital Nuernberg, Campus North, Nuremberg
  - Robert-Bosch-Hospital, Stuttgart
  - University Hospital Ulm, Ulm
- Greece (5):
  - General Hospital of Athens Laikon, Athens
  - University General Hospital "Attikon", Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patras, Pátrai
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (4):
  - Semmelweis University, Budapest
  - Szabolcs-Szatmar-Bereg County Teaching Hospital, Nyíregyháza
  - Tolna County Hospital, Szekszárd
  - Fejer County St. Gyorgy University Teaching Hospital, Székesfehérvár
- Italy (18):
  - National Hospital SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Marche University Hospital, Ancona
  - Polyclinic S. Orsola-Malpighi, Bologna
  - ASST Spedali Civili Brescia, Brescia
  - University Hospital "G.Rodolico - San Marco", Catania
  - Careggi University Hospital, Florence
  - Institute of Romagna for Cancer Research " Dino Amadori" - IRCCS IRST, Forlì
  - Maggiore Polyclinic Hospital, Foundation IRCCS Ca' Granda, Milan
  - European Institute of Oncology (IEO), IRCCS, Milan
  - University Hospital "Maggiore della Carita" of Novara, Novara
  - University Hospital San Luigi Gonzaga, Orbassano
  - University Polyclinic Hospital "Paolo Giaccone" Palermo, Palermo
  - Polyclinic San Matteo, IRCCS, Pavia
  - Local Health Company of Pesaro and Urbino, Pesaro
  - Hospital Arcispedale S. Maria Nuova of Reggio Emilia, Reggio Emilia
  - Hospital S. Eugenio- Rome 2 ASL, Rome
  - City of Health and Science of Turin, Turin
  - ASST Sette Laghi Hospital, Varese
- Poland (12):
  - "InterHem" General Partnership, Bialystok
  - University Teaching Centre, Hematology and Transplantology Clinic, Gdansk
  - Independent Public Healthcare Facility University Hospital in Krakow, Krakow
  - Nicolaus Copernicus Provincial Multispecialty Oncology and Traumatology Center, Lodz
  - Jedrzej Sniadecki Specialist Hospital in Nowy Sacz, Nowy Sącz
  - Oncology Center of Warmia and Mazury in Olsztyn, Olsztyn
  - AIDPORT, Poznan
  - Dom Lekarski Medical Center Outlet Park, Szczecin
  - Janusz Korczak Provincial Specialist Hospital, Słupsk
  - Clinical Best Solutions LLC, Limited Partnership, Warsaw
  - Dr Alfred Sokolowski Specialty Hospital, Wałbrzych
  - Jan Mikulicz-Radecki Teaching Hospital in Wroclaw, Wroclaw
- Portugal (5):
  - Hospital Center of Baixo Vouga -Aveiro Unit - Hospital Infante D. Pedro, Aveiro
  - Braga Hospital, Braga
  - Central Hospital of Western Lisbon, Lisbon
  - Centro Hospitalar Lisboa Norte (CHLN) EPE - Hospital de Santa Maria, Lisbon
  - Vila Nova de Gaia Central Hospital, Vila Nova de Gaia
- Romania (5):
  - Onco Card Srl, Brasov
  - Colentina Clinical Hospital, Department of Hematology, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Hematology Department, Cluj-Napoca
  - Bihor County Emergency Clinical Hospital, Department of Hematology, Oradea
  - Targu Mures County Emergency Clinical Hospital, Internal Medicine Department I, Hematology Unit, Târgu Mureş
- Serbia (4):
  - University Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad
- South Korea (9):
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Keimyung University - Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (12):
  - University Hospital Germans Trias i Pujol, Badalona
  - University Hospital Vall d'Hebron, Barcelona
  - Catalan Institute of Oncology, Hospital Duran i Reynals, Barcelona
  - Caceres Hospital Complex - San Pedro de Alcantara General Hospital, Cáceres
  - Gran Canaria Dr Negrin University Hospital, Las Palmas de Gran Canaria
  - University Hospital 12 de Octubre, Madrid
  - University Hospital Ramon y Cajal, Madrid
  - University Hospital Virgen de la Victoria, Málaga
  - University Clinical Hospital of Salamanca, Salamanca
  - University Clinical Hospital of Valencia, Valencia
  - University and Polytechnic Hospital La Fe, Valencia
  - Quironsalud Zaragoza Hospital, Zaragoza
- United Kingdom (14):
  - Birmingham Heartlands Hospital, Birmingham
  - Lincoln County Hospital, Boston
  - Pilgrim Hospital, Boston
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Western General Hospital, Lothian Health Board, Edinburgh
  - Gloucestershire Royal Hospital, Gloucester
  - Harrogate District Hospital, Harrogate
  - Leicester Royal Infirmary, Leicester
  - The Clatterbridge Cancer Center NHS Foundation Trust, Liverpool
  - University College Hospital, London
  - Guy's Hospital, London
  - Genesis Care, Oxford, Oxford
  - Genesis Care, Windsor, Windsor